CLINICAL TRIAL: NCT07185282
Title: A Multicenter, Randomized, Double-Blind, Vehicle-Controlled Phase 3 Study to Evaluate the Efficacy and Safety of MH004 Ointment Followed by a 44-week Open-Label Long-Term Safety Extension Period in Adolescents and Adults With Mild to Moderate Atopic Dermatitis
Brief Title: A Phase 3 Study of MH004 Ointment in Patients With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Minghui Pharmaceutical (Hangzhou) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MH004-P-302
Record Dates: First submitted 2025-09-12; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VC Period: MH004 1.0% Ointment BID (Experimental): Participants received MH004 1.0% Ointment twice daily (BID) from Day 1 to Week 8 during the Vehicle Control (VC) Period.
  Interventions: Drug: MH004 Ointment
- VC Period: Vehicle Ointment BID (Placebo Comparator): Participants received vehicle ointment BID from Day 1 to Week 8 during the VC Period.
  Interventions: Drug: Vehicle Ointment
- LTS Period: MH004 1.0% Ointment BID (Experimental): Participants who applied MH004 1.0% ointment during VC Period, continued applying MH004 1.0% ointment BID from Week 8 to 52 during the LTS Period.
  Interventions: Drug: MH004 Ointment
- LTS Period: Vehicle Ointment to MH004 1.0% Ointment BID (Placebo Comparator): Participants who applied vehicle ointment BID during the VC Period, were randomized to apply MH004 1.0% ointment topically BID from Week 8 to 52 during the LTS Period.
  Interventions: Drug: Vehicle Ointment

INTERVENTIONS:
Drug: MH004 Ointment — MH004 1% ointment applied topically to the affected area as a thin film twice daily.
  Arms: LTS Period: MH004 1.0% Ointment BID; VC Period: MH004 1.0% Ointment BID
Drug: Vehicle Ointment — Matching vehicle ointment applied topically to the affected area as a thin film twice daily.
  Arms: LTS Period: Vehicle Ointment to MH004 1.0% Ointment BID; VC Period: Vehicle Ointment BID

SUMMARY:
This is a multicenter, randomized, double-blind, vehicle-controlled phase III study of MH004 Ointment with a 44-week open-label long-term safety extension period. The study was designed to evaluate the safety, tolerability, pharmacokinetics (PK), and primary efficacy of MH004 Ointment in adolescents and adults with mild to moderate atopic dermatitis.

DETAILED DESCRIPTION:
This phase III trial of MH004 Ointment comprises two periods: a vehicle control period and an open-label long-term safety extension period. Participants will be randomly aligned to the 1.0% MH004 Ointment BID or Vehicle BID arm and treated for up to 8 weeks, followed by a 44-week open-label LTS treatment period with 1.0% MH004 Ointment BID. The primary objective of this trial is to evaluate the efficacy of MH004 Ointment in adolescent and adult participants with mild to moderate atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents aged ≥ 12 to 17 years, inclusive, and men and women aged ≥18 years.
2. Clinical diagnosis of mild to moderate atopic dermatitis (AD) for at least 1 year prior to Day 1.
3. Participants meet all the following atopic dermatitis criteria:

   VC period: IGA 2 to 3, affected BSA 3% to 20% (excluding scalp) at the baseline visit.

   LTS period: IGA 0 to 4, affected BSA 0% to 20% (excluding scalp) at Week 8.
4. Participants who agree to discontinue all agents used to treat AD from screening through the final follow-up visit.
5. Participants who have at least one AD lesion not located on the hands, feet, or genitalia.
6. Willingness to avoid pregnancy or fathering of children. -

Exclusion Criteria:

1. Unstable course of AD (spontaneously improving or rapidly deteriorating) as determined by the investigator in the 4 weeks prior to baseline.
2. Concurrent conditions and history of other diseases:

   * Immunocompromised.
   * Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before Baseline.
   * Active acute bacterial, fungal, or viral skin infection within 1 week before Baseline.
   * Any other concomitant skin disorder, pigmentation, or extensive scarring that, in the opinion of the investigator, may interfere with the evaluation of AD lesions or compromise participant safety.
   * Presence of AD lesions only on the hands or feet without prior history of involvement of other classical areas of involvement such as the face or the folds.
   * Other types of eczema.
3. Clinically significant cardiac disease; new cerebral infarction within 6 months from dosing; malignancies within 5 years from dosing; low hemoglobin; severe renal disease on dialysis; liver disease.
4. Systemic corticosteroids treated within 4 weeks before dosing; immunizations or sedating antihistamines treated within 4 weeks before dosing; other topical treatments for AD within 1 week before dosing.
5. Previously received Janus kinase (JAK) inhibitors, systemic or topical.
6. Ultraviolet light therapy or prolonged exposure to UV radiation within 2 weeks before dosing.
7. Liver function tests: AST or ALT ≥ 2 × ULN; alkaline phosphatase and/or bilirubin > 1.5 × ULN.
8. Pregnant or lactating participants, or those considering pregnancy.
9. Alcohol or drug abuse. -

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving Investigator's Global Assessment treatment success (IGA-TS) at Week 4. | Baseline to week 4.
  The IGA is an overall eczema severity rating on a 5-point scale ranging from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, induration/papulation, and oozing/crusting. The IGA-TS is defined as an IGA score of 0 (clear skin) or 1 (almost clear skin) with ≥ 2 grade improvement from Baseline.
Proportion of participants achieving EASI-75 at Week 4. | Baseline to week 4.
  EASI scoring system examines 4 areas of the body and weights them for participants of at least 8 years of age. Each of the 4 body regions is assessed separately for erythema (E), induration/papulation/edema (I), excoriations (Ex), and lichenification (l) for an average degree of severity of each sign in each region. The severity strata for the EASI are as follows: 0 = clear; 0.1 to 1.0 = almost clear; 1.1 to 7.0 = mild; 7.1 to 21.0 = moderate; 21.1 to 50.0 = severe; 50.1 to 72.0 = very severe. An EASI75 responder was defined as a participant achieving 75% or greater improvement from Baseline in EASI score.

SECONDARY OUTCOMES:
Key Secondary Endpoints: Proportion of participants achieving IGA-TS at Week 8. | Baseline to week 8.
  The IGA-TS is defined as an IGA score of 0 (clear skin) or 1 (almost clear skin) with ≥ 2 grade improvement from Baseline.
Key Secondary Endpoints: Proportion of participants achieving EASI-75 at Week 8. | Baseline to week 8.
  An EASI75 responder was defined as a participant achieving 75% or greater improvement from Baseline in EASI score.
Key Secondary Endpoints: Proportion of participants with a ≥ 4-point improvement in Itch Numerical Rating Scale (INRS) from baseline to Week 4. | From pre-dose to 4 weeks after the first dose.
  The Itch NRS is a daily patient-reported measure (24-hour recall) of the worst level of itch intensity. Participants will be asked to rate the itching severity because of their AD by selecting a number from 0 (no itch) to 10 (worst imaginable itch) that best describes their worst level of itching in the past 24 hours.
Key Secondary Endpoints: Proportion of participants with a clinically meaningful (≥ 6-point) improvement in the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form-Sleep Disturbance (8b - 24-hour recall) score at Week 4 | From pre-dose to 4 weeks after the first dose.
  This assessment is self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. PROMIS Short Form - Sleep-Related Impairment (8a) collected in the evening before sleeping; PROMIS Short Form - Sleep Disturbance (8b) collected in the morning after the participant wakes up.
Key Secondary Endpoints: Proportion of participants with a clinically meaningful (≥ 6-point) improvement in the PROMIS Short Form - Sleep - Related Impairment (8a - 24-hour recall) score at Week 4. | From pre-dose to 4 weeks after the first dose.
  This assessment is self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. PROMIS Short Form - Sleep-Related Impairment (8a) collected in the evening before sleeping; PROMIS Short Form - Sleep Disturbance (8b) collected in the morning after the participant wakes up.
Incidence, Frequency, Duration and Severity of Treatment-Emergent Adverse Event (TEAE) | From the time of Informed Consent Form signing until at least 30 days after the last application of study drug (up to Week 52)
  An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or an important medical event may be considered serious when, based on appropriate medical judgment, the event may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed above. A TEAE or treatment emergent SAE is any AE or SAE either reported for first time or worsening of a pre-existing event after first dose of study drug.
Incidence of Treatment-Emergent Serious Adverse Event (SAE) and Incidence of AEs resulting discontinue medication | From the time of Informed Consent Form signing until at least 30 days after the last application of study drug (up to Week 52)
  An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or an important medical event may be considered serious when, based on appropriate medical judgment, the event may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed above. A TEAE or treatment emergent SAE is any AE or SAE either reported for first time or worsening of a pre-existing event after first dose of study drug.
Characterization of Pharmacokinetics (Ctrough) of MH004 Ointment in Participants With Mild to Moderate Atopic Dermatitis at Week 2.4.8 during the VC period and Week 12, 24, 36, 52 during the LTS period. | Baseline, Week 2, 4, 8, 12, 24, 36, 52
  Trough drug concentration (Ctrough)
Change From Baseline in DLQI/CDLQI at Week 2, 4, 8, 12, 24, 52 | Baseline, Week 2, 4, 8, 12, 24, 52
  The DLQI/CDLQI (Dermatology Life Quality Index/Children Dermatology Life Quality Index) is a standardized tool for assessing the impact of skin diseases on patients' quality of life. It consists of 10 questions covering multiple dimensions such as symptom perception, daily activities, and social psychology. The total score ranges from 0 to 30, with a higher score indicating a more severe impact of the disease on life.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No